CLINICAL TRIAL: NCT06342180
Title: Serum Uric Acid Levels in Polycystic Ovary Syndrome Subtypes.
Brief Title: Metabolic Differences Between Subtypes of Polycystic Ovary Syndrome
Status: Completed | Type: Observational
Sponsor: Uşak University (Other)
Responsible Party: Principal Investigator, Cevdet Duran, Prof. of medicine, Uşak University
Other Study IDs: Usakupcos1
Record Dates: First submitted 2024-03-26; First posted 2024-04-02 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2024-03

CONDITIONS: Uric Acid Concentration, Serum, Quantitative Trait Locus 7; Polycystic Ovary Syndrome
Keywords: polycystic ovary syndrome; uric acid level; PCOS Subtypes
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — An amount of 2-3 ml of blood sample will be collected from the patients after 8-12 hours of fasting and will be kept frozen at -70 degrees to calculate the serum UA levels.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Controls: Healthy controls between aged 18 and 35 years
  Interventions: Diagnostic Test: Serum uric acid level
- PCOS Subtype 1: Hyperandrogenemia+oligoanovulation+PCO appearance on USG
  Interventions: Diagnostic Test: Serum uric acid level
- PCOS Subtype 2: Hyperandrogenemia+oligoanovulation
  Interventions: Diagnostic Test: Serum uric acid level
- PCOS Subtype 3: Hyperandrogenemia+ PCO appearance on USG
  Interventions: Diagnostic Test: Serum uric acid level
- PCOS Subtype 4: Oligoanovulation+ PCO appearance on USG
  Interventions: Diagnostic Test: Serum uric acid level

INTERVENTIONS:
Diagnostic Test: Serum uric acid level — An amount of 2-3 ml of blood sample will be collected from the patients after 8-12 hours of fasting and will be kept frozen at -70 degrees to calculate the serum UA level.

SUMMARY:
We aimed to investigate serum uric acid levels in patients with different phenotype of policystic ovary syndrome and to compare healthy controls.

DETAILED DESCRIPTION:
The final breakdown product of adenosine and guanosine-based purines formed as a result of the breakdown of nucleic acids is uric acid (UA). Uric acid has many beneficial and harmful properties for humans. One of the most important benefits of uric acid is that it can act as an antioxidant and is perhaps one of the most important antioxidants in plasma. However, this hypothesis is completely opposite to the hypothesis advocating an increase in the incidence of hyperuricemia and cardiovascular events. There are also experimental studies showing that UA, which has an antioxidant effect in the extracellular fluid, has harmful effects when it enters the cell. Uric acid can contribute to molecular endothelial dysfunction, oxidative stress and the formation of many oxygen radicals, disruption of the vasodilation mechanism, and increased inflammation. A correlation has been found between insulin resistance and serum UA level in patients with metabolic syndrome. It has been reported in some studies that hyperuricemia can be considered as an indicator of insulin resistance in these patients. At the same time, many studies have reported that both insulin resistance and hyperuricemia increase cardiovascular risk. In a study, it was stated that every 1 mg/dL increase in serum UA level in women increased the risk of ischemic heart disease by 12%.

Polycystic ovary syndrome (PCOS) is one of the endocrinological diseases that affects 5-20% of women of reproductive age. It is characterized by oligoanovulation, clinical or biochemical hyperandrogenemia and the appearance of polycystic ovaries. This syndrome is diagnosed according to the revised 2003 Rotterdan criteria; These criteria; 1) Oligo-anovulation, 2) Clinical and/or biochemical hyperandrogenism findings, 3) Polycystic ovary (PCO) appearance in the ovaries. For diagnosis, it is sufficient to have two of these criteria and not have another disease that causes this.

Polycystic ovary syndrome; Metabolic disorders such as insulin resistance, dyslipidemia, glucose intolerance, hypertension and obesity are often accompanied, and increased inflammation is one of the main characteristics of this syndrome. While the presence or absence of PCOS was important until recently, recent studies have shown that metabolic changes and inflammation occur at different degrees in different subtypes of PCOS. Therefore, PCOS cases are divided into 4 subtypes. These; Subtype 1 has hyperandrogenemia + oligoanovulation + PCO appearance on ultrasonography (USG), Subtype 2 has hyperandrogenemia + oligoanovulation, Subtype 3 has hyperandrogenemia + PCO appearance on USG, and Subtype 4 has oligoanovulation + PCO appearance on USG. As the subtype number of polycystic ovary syndrome decreases, the severity and frequency of metabolic disorders and inflammation accompanying polycystic ovary syndrome increase.

Hyperuricemia is one of the common metabolic disorders in patients with PCOS. Prevalence studies have shown that the frequency of hyperuricemia in patients with PCOS is approximately 25%, 3 times higher than in controls. However, these studies were conducted in the general PCOS patient group, and patients with different subtypes were not evaluated.

Since there are different metabolic effects in different subtypes of polycystic ovary syndrome; In this study we aimed to investigate whether there is a difference between serum UA levels in different PCOS subtypes. Studies investigating UA levels in subtypes of PCOS are rare in the literature. We aim to contribute to the knowledge in this field with the results we obtained from this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who applied for reasons such as hair growth, acne, menstrual irregularity or infertility and were diagnosed with PCOS after examination, biochemical, hormonal and sonographic tests,
2. Female patients between the ages of 18-35,
3. Patients without known cancer, liver or kidney failure,
4. Patients who do not take medications that will affect uric acid levels,
5. Female patients without active infection will be included. -

Exclusion Criteria:

1. Female patients under eighteen years of age and >35 years of age,
2. Patients with known cancer, liver and kidney failure,
3. Patients taking medications that will affect uric acid levels,
4. Patients with active infection will be excluded. -

Ages: 18 Years to 35 Years | Sex: Female
Age Groups: Adult
Study Population: Women aged between 18 and 35, age-matched between groups, diagnosed with PCOS and without a known cancer diagnosis, liver and kidney failure, not taking medications that would affect uric acid levels, and without active infection.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Uric acid levels in PCOS subtypes | Eight months
  Since there are different metabolic effects in different subtypes of polycystic ovary syndrome; In this study we aimed to investigate whether there is a difference between serum UA levels in different PCOS subtypes and the difference between these subtypes and the healthy group.

CONTACTS AND LOCATIONS:
Locations (1):
- Usak Egitim Ve Araştırma Hastanesi, Uşak, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided